CLINICAL TRIAL: NCT00032344
Title: CSP #380 - Prospective Evaluation of Risk Factors for Large (> 1 CM) Colonic Adenomas in Asymptomatic Subjects
Brief Title: Long-term Follow-up Study Designed to Evaluate the Relative Risk of Two Colonoscopy Schedules for Patients With Small Polyps
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Lieberman, David - Study Chair, Department of Veterans Affairs
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 380
Record Dates: First submitted 2002-03-18; First posted 2002-03-19 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Colorectal Cancer
Keywords: large (>1 cm) adenomas
MeSH Terms: conditions — Colorectal Neoplasms; Adenoma | interventions — Colonoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Other): Phase I - Cross-sectional; Phase II - 5 year follow-up; Phase III - 10 year follow-up
  Interventions: Procedure: Colonoscopy

INTERVENTIONS:
Procedure: Colonoscopy — Phase I - Cross-sectional; Phase II - 5 year follow-up; Phase III - 10 year follow-up

SUMMARY:
Colorectal cancer is a leading cause of cancer death in the United States. Mortality remains high because most colorectal cancers are detected after there has been regional or distant spread, precluding curative surgical resection. With this in mind, screening strategies have been recommended for asymptomatic individuals which hope to reduce mortality from colon cancer by detecting and removing premalignant adenomatous polyps or early malignant lesions. Screening of asymptomatic individuals over age 50 with sigmoidoscopy and fecal occult blood tests has been advocated by the American Cancer Society. However, current screening will identify only 50% of patients who have adenomatous polyps. More sensitive tests for polyp detection, like colonoscopy, are costly, require extensive resources and are unlikely to be used for screening large populations. Ideal screening would identify patients with the highest risk of cancer and target more sensitive screening tests at this population. The identification of low cost, easily collectible risk factors which can be used to target patients for the more sensitive screening tests is the primary purpose of this study. Since a major segment of the veteran population is over the age of 50, there will be a substantial impact in reduction of both mortality and morbidity due to colon cancer and attendant cost savings to the VA for treatment if such risk factors can be identified.

Phase I is a cross-sectional study designed to identify risk factors for large (>1 cm) adenomatous polyps. Approximately 3200 asymptomatic subjects (age 50-75) have completed risk factor assessment, medical and dietary histories, and have undergone complete colonoscopy examination. This will identify for comparison purposes a polyp-free control group and is the first large prospective study to include such a group. Data at colonoscopy will characterize the prevalence, size and distribution of adenomatous polyps. This will permit an assessment of sensitivity of sigmoidoscopy in this population. In addition, tissue from normal rectal mucosa will be analyzed for evidence of cell proliferation activity. The primary focus of Phase I is a risk factor analysis. A multivariate analysis will be performed to determine the relationship of historical and environmental factors as well as cell proliferation activity with the presence of adenomatous polyps. A cohort consisting of a subgroup of polyp patients (large and small) and matched polyp-free controls will be tracked longitudinally to determine polyp occurrence/recurrence rates.

Phase II of the study is a long-term follow-up study designed to evaluate the relative risk of two repeat colonoscopies.

Phase III is an extension in follow-up of an additional five years, a total of ten years in all, to include all study patients. The primary focus will be on documenting long-term mortality and medical outcomes as well as occurrence/reoccurrence of neoplasia with special emphasis on ten-year cancer rates.

DETAILED DESCRIPTION:
Primary Hypothesis: Risk factors can be determined for large (>1 cm) adenomas, precursor lesions for colorectal cancer.

Secondary Hypothesis: Determine long-term rates for development or recurrence of polyps; determine sensitivity/specificity of current colon cancer screening strategies; determine relationship of dietary factors and biomarkers of cell proliferation; determine the efficacy and safety of long-term (5 years) repeat colonoscopy in patients with small polyps.

Intervention: Phase I: All patients undergo full colonoscopy. Phase II: Randomization to repeat colonoscopy at 2-3 years and 5 years after baseline, or, repeat colonoscopy at 5 years only. Phase III: Ten-year follow-up on all Phase I patients for medical outcomes. Repeat colonoscopy at 10 years on polyp-free patients (Phase I) aged 50-64.

Primary Outcomes: Presence of risk factors and adenomatous polyps including prevalence, descriptive characteristics, and long-term occurrence/recurrence rates.

Study Abstract: Phase I is a cross-sectional study designed to identify risk factors for large (>1 cm) adenomatous polyps. Approximately 3200 asymptomatic subjects (age 50-75) have completed risk factor assessment, medical and dietary histories, and have undergone complete colonoscopy examination. This will identify for comparison purposes a polyp-free control group and is the first large prospective study to include such a group. Data at colonoscopy will characterize the prevalence, size and distribution of adenomatous polyps. This will permit an assessment of sensitivity of sigmoidoscopy in this population. In addition, tissue from normal rectal mucosa will be analyzed for evidence of cell proliferation activity. The primary focus of Phase I is a risk factor analysis. A multivariate analysis will be performed to determine the relationship of historical and environmental factors as well as cell proliferation activity with the presence of adenomatous polyps. A cohort consisting of a subgroup of polyp patients (large and small) and matched polyp-free controls will be tracked longitudinally to determine polyp occurrence/recurrence rates.

Phase II of the study is a long-term follow-up study designed to evaluate the relative risk of two repeat colonoscopy schedules for patients with small polyps identified in Phase I of the study. Recruitment is complete with 615 patients eligible (of the target 808) assigned at random to either repeat colonoscopy at 2-3 years and 5 years, or to repeat colonoscopy at 5 years only. This phase will also provide preliminary longitudinal risk factor information related to occurrence/recurrence of polyps.

Phase III was a 5-year extension of follow-up period. All Phase I patients were to be reconsented to provide medical outcome data for a period of 10 years from baseline exam. Phase I patients polyp-free, aged 50-64 will be offered repeat colonoscopy at 10 years to evaluate long-term risk.

Results (Phase I): 3121 patients had complete colonoscopy which revealed high rates of neoplasia: 37.5% had one or more neoplastic lesions; 10.5% had advanced neoplasia including 30 cases of invasive cancer (1%). There were 3.7% of patients with no lesions in the rectum or sigmoid colon who had advanced neoplasia elsewhere in the colon: 32% of all patients with advanced neoplasia would not be detected with an exam of the rectum or sigmoid colon (distal); 62% of patients with proximal advanced neoplasia would not be detected with an exam of the rectum and sigmoid colon. There were few serious complications (0.3%).

The one-time fecal occult blood test (FOBT) was evaluated as a diagnostic test for advanced neoplasia. A positive FOBT indicated an increased likelihood (3-4x) of advanced neoplasia. However, one-time FOBT failed to detect 75% of patients with advanced neoplasia.

The primary analysis of risk factors (Phase I) found positive associations (for advanced neoplasia) for history of a first degree relative with colorectal cancer (OR, 1.66; 95% CI, 1.16-2.35), current smoking (OR, 1.85; 95% CI, 1.33-2.58), and current moderate to heavy alcohol use (OR, 1.02, 95% CI, 1.01-1.03). Inverse associations were found for cereal fiber intake (OR, 0.95, 95% CI, 0.91-0.99), vitamin D intake (OR, 0.94, 95% CI, 0.90-0.99), and use of NSAIDs (OR, 0.66, 95% CI, 0.48-0.91). Results appeared in JAMA (2003;290:2959-2967).

Phase III is completed with patients completing their scheduled follow-ups. A major manuscript on the sensitivity/specificity of digital rectal exam appeared in Annals of Internal Medicine January, 2005. The Phase II results manuscript appeared in Gastroenterology in October 2007.

ELIGIBILITY:
Inclusion Criteria:

Study Complete

Exclusion Criteria:

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3200 (Actual)
Dates: Start 1993-10; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Phase I: Risk factors include: family history; dietary; fat, fiber, calcium; alcohol history; tobacco use; physical activity; obesity; NSAID use; and, biomarkers: BRDU, PCNA | Cross-sectional

SECONDARY OUTCOMES:
Phase II: Colonoscopy outcomes to determine recurrence rates and compare surveillance strategies | 5 years
Phase III: Medical outcomes including mortality. Colonoscopy outcomes in subgroup of polyp free patient at baseline to determine long term risk. | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: David Lieberman, MD, Study Chair — VA Medical Center, Portland
Locations (13):
- United States (13):
  - Carl T. Hayden VA Medical Center, Phoenix, Arizona
  - Southern Arizona VA Health Care System, Tucson, Tucson, Arizona
  - VA Medical Center, Long Beach, Long Beach, California
  - VA Palo Alto Health Care System, Palo Alto, California
  - VA Medical Center, San Francisco, San Francisco, California
  - VA Eastern Colorado Health Care System, Denver, Denver, Colorado
  - Edward Hines, Jr. VA Hospital, Hines, Illinois
  - VA Medical Center, Minneapolis, Minneapolis, Minnesota
  - VA Medical Center, Kansas City MO, Kansas City, Missouri
  - VA Medical Center, Durham, Durham, North Carolina
  - VA Medical Center, Portland, Portland, Oregon
  - VA North Texas Health Care System, Dallas, Dallas, Texas
  - VA Medical & Regional Office Center, White River, White River Junction, Vermont

REFERENCES:
- [Result] Schreiner MA, Weiss DG, Lieberman DA. Proximal and large hyperplastic and nondysplastic serrated polyps detected by colonoscopy are associated with neoplasia. Gastroenterology. 2010 Nov;139(5):1497-502. doi: 10.1053/j.gastro.2010.06.074. Epub 2010 Jul 13. PMID 20633561